CLINICAL TRIAL: NCT07338812
Title: Efficacy of Virtual Reality and Whole Body Vibration on Muscle Strength and Balance in Children With Duchenne Muscular Dystrophy
Brief Title: Virtual Reality and Whole Body Vibration on Muscle Strength and Balance in Children With DMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa S Ali, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006030
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Virtual reality; whole-body vibration; muscle strength; balance; children; Duchenne muscular dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (Experimental): group (A) had designed physical therapy in addition to virtual reality
  Interventions: Device: virtual reality
- whole-body vibration (Experimental): group (B) had the same physical therapy program with whole-body vibration
  Interventions: Device: whole body vibration

INTERVENTIONS:
Device: virtual reality — Group (A) had designed physical therapy in form of Warm up with gentle stretching movements to prevent injuries. The lower limb muscles on both sides were stretched for 20 seconds, followed by 20 seconds of relaxation, five times. The quadriceps, hamstrings, anterior tibial group, calf muscles, biceps, and triceps were also contracted isometrically. Every muscle contraction was held for 5 seconds, followed by 5 seconds of relaxation, and the process was repeated five times in addition to virtual reality inform of VR program. Nintendo Wii Fit Balance Board (Nintendo, Kyoto, Japan) was used to perform the exercises. In each session, VR was used for a total of 10 minutes three times per week for three consecutive months.
  Arms: virtual reality
Device: whole body vibration — Group (B) had the same physical therapy program with WBV (Power Plate Pro 5) for a total of 10 minutes per session. The apparatus was set at 30 Hz frequency, 2 mm amplitude, and 5 minutes of operating time. The children were squatted down completely on a vibrating, side-alternating platform and were told to stay that way throughout the experience, communicating any pain they felt to the researchers. The vibration feature automatically shuts off after 5 minutes. After that, the children took a one-minute break. Then, with the same settings as those used in the squatting position, children stood on the vibration platform for 5 minutes. In each session, WBV was used for a total of 10 minutes three times per week for three consecutive months.
  Arms: whole-body vibration

SUMMARY:
we measure balance and quadriceps strength in Duchenne muscular dystrophy children after applying virtual reality and whole body vibration

DETAILED DESCRIPTION:
Two groups of fifty children with Duchenne muscular dystrophy, aged 6 to 10, were randomly assigned after being selected from the outpatient clinic of faculty of physical therapy, Cairo University. Both groups (A and B) participated in physical treatment for three consecutive months; group (A) had designed physical therapy in addition to virtual reality, whereas group (B) had the same physical therapy program with whole-body vibration three times per week.

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed with DMD
* aged between 6 and 10 years
* having lower extremities and trunk muscle strength of grade 3+
* were able to move their upper and lower limbs normally and being able to walk unhindered at levels I and II of the Ambulation function classification system for DMD (AFCSD)

Exclusion Criteria:

* cardiopulmonary dysfunction or skeletal abnormalities that are either congenital or acquired
* had previously experienced lower limb surgical procedure
* had neurological conditions that affected their balance and gait or had poor motor development
* exhibited behavioural disorders preventing them from cooperating during the trial
* being overweight (body mass index (BMI) >25 kg/ m2) because a lot of fat makes it hard for the ultrasound to measure thickness

Ages: 6 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — muscular dystrophy predominantly affecting boys
Enrollment: 50 (Actual)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-10-12 (Actual)

PRIMARY OUTCOMES:
balance | 12 weeks
  Biodex Balance System (BBS) (BSS; Biodex, Inc, Shirley, NY) was used to evaluate each child's dynamic balance. It is a multiaxial tool that records and evaluates a person's capacity to maintain joint stability under dynamic stress. The BBS uses a circular platform that can move concurrently in the anterior-posterior and medial-lateral axes, unlike force plate technologies.
quadriceps muscle strength | 12 weeks
  The Lafayette Manual Muscle Tester (MMT) Model Number 01163 combines accuracy and precision with contemporary ergonomic design to generate exact, impartial, and reliable results. The three replaceable, cushioned stirrups made it possible to employ established methods with assurance and effectiveness while preserving patient comfort

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo university, Cairo
  - Cairo university, Giza

IPD SHARING:
Plan to Share IPD: Undecided